CLINICAL TRIAL: NCT04032379
Title: Diagnostic and Prognostic Biomarkers of Idiopathic Intracranial Hypertension
Status: Recruiting | Type: Observational
Sponsor: Danish Headache Center (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Johanne Severinsen, Clinical assistant, M.D., Danish Headache Center
Other Study IDs: S-20170058
Record Dates: First submitted 2019-07-12; First posted 2019-07-25 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Benign Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Plasma Serum Cerebrospinalfluid (supernatant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Certain IIH or IIH-WOP: According to revised diagnostic criteria, Friedmann, 2013.
  Interventions: Other: Standard treatment
- Suspected IIH: IIH is suspected, does not fulfill diagnostic criteria.
  Interventions: Other: Standard treatment
- IIH ruled out: Patients in whom another diagnosis is made.
  Interventions: Other: Standard treatment

INTERVENTIONS:
Other: Standard treatment — No intervention, some patients have additional neuro-psychological testing.

SUMMARY:
Idiopathic intracranial hypertension (IIH) is a condition of unknown etiology, primarily affecting overweight females of childbearing age. Typically, patients experience headache and visual symptoms due to increased intracranial pressure (ICP) and papilledema. The diagnosis is difficult, and outcomes vary from no sequelae to blindness or chronic headaches. No clear prognostic indicators exist. Treatment consists of medication, weight loss, and possibly surgical intervention.There is an unmet need of defining biomarkers with prognostic or diagnostic value and defining predictors of a poor outcome.

This project is a prospective, population-based cohort study including clinical data and a biobank (blood samples and cerebrospinal fluid).

The investigator's primary aim is to identify biomarkers of diagnostic or prognostic value and to create a clinical IIH database. The clinical database will answer questions about patient characteristics at baseline and during follow-up, identify predictors of outcome, and help create a standardized programme for follow-up and

DETAILED DESCRIPTION:
This study is a multicenter, prospective, population-based cohort study with consecutive inclusion of patients in which the diagnosis of IIH is suspected. This study is carried out in collaboration between the Danish Headache Center, Rigshospitalet-Glostrup, and the Neurological Department at Odense University Hospital.

Patients are eligible for inclusion into the study if:

1. IIH is suspected
2. > 18 years old and able to provide written informed consent.

At baseline included patients will have:

A.) Medical history B.) Neurological, ophthalmological and general medical examination C.) Relevant neuro-imaging D.) Blood samples and lumbar puncture F.) Evaluation by other specialist, including neuro-psychologists, if appropriate.

Subsequently patients are divided into three sub-groups according to revised Friedmann criteria:

1. Certain IIH or IIH-WOP
2. Suspected, but unconfirmed, IIH
3. IIH ruled out

Patients are followed at a headache center and by neuro-ophthalmologist according to standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Able to and willing to provide informed consent
2. More than 18 years of age
3. Suspicion of IIH (based on clinical evaluation by neurologist or opthalmologist)

Exclusion Criteria:

1.) Unable to consent (e.g. language, mental retardation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All admitted or out-patient referrals where IIH is suspected. Patients will be identified and included consecutively once there is a clinical suspicion of IIH, if they wish to participate. Most often IIH will be suspected in a typical patient (female, child-bearing age, overweight) with either bilateral papiledema and normal neuro-imaging, high ICP by lumbar puncture or a new headache with associated visual disturbances or pulsatile tinnitus.
  All hospitals in the Capital Region of Denmark and the Southern Region of Denmark can participate and refer patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-14 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of IIH (diagnostic and prognostic) | 2 years
  Analyses of CSF and blood for protein-markers (method: Proteomics)
Visual status at conclusion of study | 2 years
  Assessment of visual fields
Visual status at conclusion of study | 2 years
  Assessment of OCT
Visual status at conclusion of study | 2 years
  Assessment of visual acuity
Headache status at conclusion of study | 2 years
  Prevalence of chronic headache (>=15 headache days per month)
Biomarkers of IIH (diagnostic and prognostic) | 2 years
  Analyses of CSF and blood for markers of metabolism (method: Metabolomics)

SECONDARY OUTCOMES:
Baseline characteristics related to poor outcome | 1 year
  Poor outcome is defined as either a.) Persistent visual field defects, decreased visual acuity after 12 months and or b.) Headache >= 15 days per month after 12 months
Results of neuropsychological evaluations | 1 year
  Standard neuro-psychological tests
Treatment and follow-up | 3 years
  Length and type of treatment and follow-up
Baseline characteristics related to IIH diagnosis | 2 years
  Evaluation of disease presentation in the different sub-groups focusing on headache phenotype, visual disturbances and pulsatile tinnitus.
Weight change in a standard care program | 2 years
  Unit of measurement is BMI
Diagnostic criteria and their use in the clinical setting | 2 years
  Revised Friedmann criteria of 2013
Clinical markers related to disease activity | 2 years
  Clinical markers of relevance: Headache phenotype, pulsatile tinnitus, visual disturbances, weight changes.
Development of IIH or IIHWOP in patients with borderline elevated ICP not fulfilling diagnostic criteria at baseline | 2 years
  ICP is measured by lumbar puncture, borderline elevated ICP is considered >20-30 mmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Rigmor Jensen, M.D., Dr.Med., Study Director — The Danish Headache Center, Rigshospitalet-Glostrup; Dagmar Beier, M.D., Ph.D., Study Director — Odense University Hospital
Locations (2):
- Denmark (2):
  - The Danish Headache Center, Department of Neurology, Rigshospitalet-Glostrup, Copenhagen, Glostrup
  - Odense University Hospital, Department of Neurology, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Durcan FJ, Corbett JJ, Wall M. The incidence of pseudotumor cerebri. Population studies in Iowa and Louisiana. Arch Neurol. 1988 Aug;45(8):875-7. doi: 10.1001/archneur.1988.00520320065016. PMID 3395261
- [Background] Wall M, Kupersmith MJ, Kieburtz KD, Corbett JJ, Feldon SE, Friedman DI, Katz DM, Keltner JL, Schron EB, McDermott MP; NORDIC Idiopathic Intracranial Hypertension Study Group. The idiopathic intracranial hypertension treatment trial: clinical profile at baseline. JAMA Neurol. 2014 Jun;71(6):693-701. doi: 10.1001/jamaneurol.2014.133. PMID 24756302
- [Background] Yri HM, Jensen RH. Idiopathic intracranial hypertension: Clinical nosography and field-testing of the ICHD diagnostic criteria. A case-control study. Cephalalgia. 2015 Jun;35(7):553-62. doi: 10.1177/0333102414550109. Epub 2014 Sep 16. PMID 25228684
- [Background] Yri HM, Ronnback C, Wegener M, Hamann S, Jensen RH. The course of headache in idiopathic intracranial hypertension: a 12-month prospective follow-up study. Eur J Neurol. 2014 Dec;21(12):1458-64. doi: 10.1111/ene.12512. Epub 2014 Jul 29. PMID 25070715
- [Background] Yri HM, Fagerlund B, Forchhammer HB, Jensen RH. Cognitive function in idiopathic intracranial hypertension: a prospective case-control study. BMJ Open. 2014 Apr 8;4(4):e004376. doi: 10.1136/bmjopen-2013-004376. PMID 24713214
- [Background] Digre KB, Nakamoto BK, Warner JE, Langeberg WJ, Baggaley SK, Katz BJ. A comparison of idiopathic intracranial hypertension with and without papilledema. Headache. 2009 Feb;49(2):185-93. doi: 10.1111/j.1526-4610.2008.01324.x. PMID 19222592
- [Background] Peng KP, Fuh JL, Wang SJ. High-pressure headaches: idiopathic intracranial hypertension and its mimics. Nat Rev Neurol. 2012 Dec;8(12):700-10. doi: 10.1038/nrneurol.2012.223. Epub 2012 Nov 20. PMID 23165338
- [Background] Headache Classification Committee of the International Headache Society (IHS). The International Classification of Headache Disorders, 3rd edition (beta version). Cephalalgia. 2013 Jul;33(9):629-808. doi: 10.1177/0333102413485658. No abstract available. PMID 23771276
- [Background] Nielsen HH, Beck HC, Kristensen LP, Burton M, Csepany T, Simo M, Dioszeghy P, Sejbaek T, Grebing M, Heegaard NH, Illes Z. The Urine Proteome Profile Is Different in Neuromyelitis Optica Compared to Multiple Sclerosis: A Clinical Proteome Study. PLoS One. 2015 Oct 13;10(10):e0139659. doi: 10.1371/journal.pone.0139659. eCollection 2015. PMID 26460890
- [Derived] Hansen NS, Korsbaek JJ, Yri HM, Jensen RH, Beier D. Are the ICHD-3 criteria for headache attributed to idiopathic intracranial hypertension valid? Headache phenotyping and field-testing in newly diagnosed idiopathic intracranial hypertension. Cephalalgia. 2024 Apr;44(4):3331024241248210. doi: 10.1177/03331024241248210. PMID 38663903